CLINICAL TRIAL: NCT00114881
Title: Urban Environment and Childhood Asthma (URECA)
Brief Title: Urban Environmental Factors and Childhood Asthma
Acronym: URECA
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Inner-City Asthma Consortium (Network); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DAIT ICAC-07; NIAID CRMS ID#: 20126 (Other: DAIT NIAID)
Record Dates: First submitted 2005-06-17; First posted 2005-06-20 (Estimated); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Asthma; Allergy
Keywords: Children; Urban Health; Pregnancy; Asthma
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Sample of umbilical cord blood (mother)
  * Maternal blood sample
  * Blood and nasal mucus collection (infant through age 14 or 16 years)
  * DNA sample of mother and child
  * Urine sample
  * Saliva sample
  * Nasal epithelial cells sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Inner-city children with asthma: Children at high risk for developing allergic diseases and asthma, on the basis of a parental history of asthma, allergic rhinitis or atopic dermatitis, and residence in the inner city

SUMMARY:
Minority children who grow up in poor urban neighborhoods have the highest rates of asthma, and also experience greater morbidity from acute exacerbations of this disease. The aim of this study is to further identify environmental factors unique to the inner city that affect immune development and the expression of wheezing, atopy and asthma for purposes of identifying new strategies for asthma prevention.

DETAILED DESCRIPTION:
The purpose of this study is to determine the way environmental factors (like the components of inner-city household dust) affect immune system development and symptoms of asthma in inner city children. The study is divided into five periods, as the subjects age from birth to 17 years old. Each age bracket will explore different objectives and endpoints.

Study Objectives/Hypotheses:

1. Subjects age 0 to 3 years old:

   * Environmental factors in the inner city adversely influence the development of the immune system to promote cytokine dysregulation, allergy, and recurrent wheezing by age 3.
   * Children who have had a viral lower respiratory infection and have developed cytokine dysregulation by age 3 are at increased risk for the development of asthma by age 6.
2. Subjects age 4 to 7 years old:

   * There is a unique pattern of immune development that is driven by specific urban exposures in early life, and this pattern of immune development is characterized by: 1) impairment of antiviral responses and 2) accentuation of Th2-like responses (e.g. cockroach-specific Interleukin-13(IL-13)). The clinical effects of these changes in immune development are frequent virus-induced wheezing and allergic sensitization by 3-4 years of age, and these characteristics synergistically increase the risk of asthma at age 7 years.
3. Subjects age 7 to 10 years old:

   * There are unique combinations of environmental exposures (cockroach allergens, indoor pollutants [Environmental Tobacco Smoke (ETS) and Nitrogen Dioxide (NO2)], lack of microbial exposure), and family characteristics (stress, genetic factors related to innate immunity) that synergistically promote asthma onset, persistence, and morbidity in urban neighborhoods. These exposures and characteristics influence immune expression and lung development during critical periods of growth, resulting in specific asthma phenotypes.
4. Subjects age 10 to 16 years old:

   -To determine the wheezing, asthma and atopy phenotypes in minority children growing up in poor urban neighborhoods as they develop from birth through adolescence.
5. Subjects to age 17 (Continuation of phase 4 to follow participants to age 17) To determine the wheezing, asthma and atopy phenotypes in minority children growing up in poor urban neighborhoods as they develop from birth through adolescence.

ELIGIBILITY:
Inclusion Criteria for Mothers:

* Plan to give birth at the study hospital
* Have asthma, hay fever, or eczema (or infant's father has any of these diseases)
* Currently reside in a pre-selected area containing at least 20% of households below the U.S. government poverty level
* At least 34 weeks pregnant at time of delivery
* Willing to allow an umbilical cord blood specimen to be obtained from her infant
* Willing to comply with all study requirements
* Have access to a phone
* Speak English. Spanish-speaking participants enrolled at sites with Spanish-speaking staff are also eligible.

Exclusion Criteria for Mothers:

* HIV infected at the time of delivery
* Plan to move out of the geographic area during the study

Exclusion Criteria for Infants:

* Respiratory distress requiring intubation and ventilation for 4 hours or more
* Respiratory distress requiring either supplemental oxygen or continuous positive airway pressure (CPAP) for 4 days or more
* Pneumonia requiring antibiotic treatment for 1 week or more
* Significant congenital abnormality
* Received palivizumab for respiratory syncytial virus prophylaxis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inner city children
Sampling Method: Non-Probability Sample
Enrollment: 560 (Actual)
Dates: Start 2005-02-02 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Development of wheezing | 0 to 3 years of age
  Establish in inner city children the immunologic causes for the development of recurrent wheezing.
Correlation of Immunologic Factors and Development of Asthma | by 7 years of age
  Establish, in this cohort of inner-city children, the immunologic causes for the development of asthma at age 7
Correlation of Risk Factors to Rapidly Evolving Asthma Phenotypes | up to 10 years of age
  Fully define the rapidly evolving asthma phenotypes and further delineate the role of risk factors related to environmental exposure (e.g.; house dust levels found through home inspection), immune development, lung growth on the natural history of asthma and allergic diseases in urban minority children
Incidence of Asthma | up to 17 years of age
  Number of participants with the incidence (development) of asthma
Occurrence of Specific Phenotypes of Asthma | up to 17 years of age
  Further define asthma phenotypes based on the findings in Inner-city Asthma Consortium-19 (ICAC-19) (Asthma Phenotypes in the Inner City (APIC), ClinicalTrials.gov Identifier NCT01383941).

CONTACTS AND LOCATIONS:
Overall Officials: James E. Gern, MD, Study Chair — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - Pediatric Clinical Research Unit, Johns Hopkins University, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Saint Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York

REFERENCES:
- [Background] Lee WM, Grindle K, Pappas T, Marshall DJ, Moser MJ, Beaty EL, Shult PA, Prudent JR, Gern JE. High-throughput, sensitive, and accurate multiplex PCR-microsphere flow cytometry system for large-scale comprehensive detection of respiratory viruses. J Clin Microbiol. 2007 Aug;45(8):2626-34. doi: 10.1128/JCM.02501-06. Epub 2007 May 30. PMID 17537928
- [Background] Lee WM, Kiesner C, Pappas T, Lee I, Grindle K, Jartti T, Jakiela B, Lemanske RF Jr, Shult PA, Gern JE. A diverse group of previously unrecognized human rhinoviruses are common causes of respiratory illnesses in infants. PLoS One. 2007 Oct 3;2(10):e966. doi: 10.1371/journal.pone.0000966. PMID 17912345
- [Result] Gold DR, Bloomberg GR, Cruikshank WW, Visness CM, Schwarz J, Kattan M, O'Connor GT, Wood RA, Burger MS, Wright RJ, Witter F, Lee-Parritz A, Sperling R, Sadovsky Y, Togias A, Gern JE. Parental characteristics, somatic fetal growth, and season of birth influence innate and adaptive cord blood cytokine responses. J Allergy Clin Immunol. 2009 Nov;124(5):1078-87. doi: 10.1016/j.jaci.2009.08.021. PMID 19895995
- [Result] Zook PM, Jordan C, Adams B, Visness CM, Walter M, Pollenz K, Logan J, Tesson E, Smartt E, Chen A, D'Agostino J, Gern JE. Retention strategies and predictors of attrition in an urban pediatric asthma study. Clin Trials. 2010 Aug;7(4):400-10. doi: 10.1177/1740774510373798. Epub 2010 Jun 22. PMID 20571137
- [Result] Kakumanu S, Jaffee K, Visness CM, Dresen A, Burger M, Witter FR, O'Connor GT, Cruikshank WW, Shreffler WG, Bacharier LB, Gern JE. The influence of atopy and asthma on immune responses in inner-city adults. Immun Inflamm Dis. 2016 Feb 26;4(1):80-90. doi: 10.1002/iid3.96. eCollection 2016 Mar. PMID 27042305
- [Result] Gruenberg DA, Wright RJ, Visness CM, Jaffee KF, Bloomberg GR, Cruikshank WW, Kattan M, Sandel MT, Wood RA, Gern JE. Relation between stress and cytokine responses in inner-city mothers. Ann Allergy Asthma Immunol. 2015 Nov;115(5):439-445.e3. doi: 10.1016/j.anai.2015.07.021. Epub 2015 Sep 26. PMID 26409873
- [Result] McGowan EC, Bloomberg GR, Gergen PJ, Visness CM, Jaffee KF, Sandel M, O'Connor G, Kattan M, Gern J, Wood RA. Influence of early-life exposures on food sensitization and food allergy in an inner-city birth cohort. J Allergy Clin Immunol. 2015 Jan;135(1):171-8. doi: 10.1016/j.jaci.2014.06.033. Epub 2014 Aug 13. PMID 25129677
- [Result] Lynch SV, Wood RA, Boushey H, Bacharier LB, Bloomberg GR, Kattan M, O'Connor GT, Sandel MT, Calatroni A, Matsui E, Johnson CC, Lynn H, Visness CM, Jaffee KF, Gergen PJ, Gold DR, Wright RJ, Fujimura K, Rauch M, Busse WW, Gern JE. Effects of early-life exposure to allergens and bacteria on recurrent wheeze and atopy in urban children. J Allergy Clin Immunol. 2014 Sep;134(3):593-601.e12. doi: 10.1016/j.jaci.2014.04.018. Epub 2014 Jun 4. PMID 24908147
- [Result] Gern JE, Pappas T, Visness CM, Jaffee KF, Lemanske RF, Togias A, Bloomberg GR, Cruikshank WW, Lamm C, Tuzova M, Wood RA, Lee WM. Comparison of the etiology of viral respiratory illnesses in inner-city and suburban infants. J Infect Dis. 2012 Nov;206(9):1342-9. doi: 10.1093/infdis/jis504. Epub 2012 Sep 25. PMID 23014674
- [Result] Heymann PW, Platts-Mills TA. Deciphering the importance of host and environmental factors that influence the genesis of asthma during childhood. J Infect Dis. 2012 Nov;206(9):1331-3. doi: 10.1093/infdis/jis507. Epub 2012 Sep 25. No abstract available. PMID 23014673
- [Result] McLoughlin RM, Calatroni A, Visness CM, Wallace PK, Cruikshank WW, Tuzova M, Ly NP, Ruiz-Perez B, Kattan M, Bloomberg GR, Lederman H, Gern JE, Gold DR. Longitudinal relationship of early life immunomodulatory T cell phenotype and function to development of allergic sensitization in an urban cohort. Clin Exp Allergy. 2012 Mar;42(3):392-404. doi: 10.1111/j.1365-2222.2011.03882.x. Epub 2011 Nov 9. PMID 22092655
- [Result] Sumino K, Tucker J, Shahab M, Jaffee KF, Visness CM, Gern JE, Bloomberg GR, Holtzman MJ. Antiviral IFN-gamma responses of monocytes at birth predict respiratory tract illness in the first year of life. J Allergy Clin Immunol. 2012 May;129(5):1267-1273.e1. doi: 10.1016/j.jaci.2012.02.033. Epub 2012 Mar 27. PMID 22460071
- [Result] Chi A, Wildfire J, McLoughlin R, Wood RA, Bloomberg GR, Kattan M, Gergen P, Gold DR, Witter F, Chen T, Holick M, Visness C, Gern J, O'Connor GT. Umbilical cord plasma 25-hydroxyvitamin D concentration and immune function at birth: the Urban Environment and Childhood Asthma study. Clin Exp Allergy. 2011 Jun;41(6):842-50. doi: 10.1111/j.1365-2222.2011.03712.x. Epub 2011 Apr 11. PMID 21481021
- [Result] Wood RA, Bloomberg GR, Kattan M, Conroy K, Sandel MT, Dresen A, Gergen PJ, Gold DR, Schwarz JC, Visness CM, Gern JE. Relationships among environmental exposures, cord blood cytokine responses, allergy, and wheeze at 1 year of age in an inner-city birth cohort (Urban Environment and Childhood Asthma study). J Allergy Clin Immunol. 2011 Apr;127(4):913-9.e1-6. doi: 10.1016/j.jaci.2010.12.1122. Epub 2011 Feb 18. PMID 21333343
- [Result] Gern JE. The Urban Environment and Childhood Asthma study. J Allergy Clin Immunol. 2010 Mar;125(3):545-9. doi: 10.1016/j.jaci.2010.01.037. PMID 20226291
- [Result] Wright RJ, Visness CM, Calatroni A, Grayson MH, Gold DR, Sandel MT, Lee-Parritz A, Wood RA, Kattan M, Bloomberg GR, Burger M, Togias A, Witter FR, Sperling RS, Sadovsky Y, Gern JE. Prenatal maternal stress and cord blood innate and adaptive cytokine responses in an inner-city cohort. Am J Respir Crit Care Med. 2010 Jul 1;182(1):25-33. doi: 10.1164/rccm.200904-0637OC. Epub 2010 Mar 1. PMID 20194818
- [Result] Gern JE, Visness CM, Gergen PJ, Wood RA, Bloomberg GR, O'Connor GT, Kattan M, Sampson HA, Witter FR, Sandel MT, Shreffler WG, Wright RJ, Arbes SJ Jr, Busse WW. The Urban Environment and Childhood Asthma (URECA) birth cohort study: design, methods, and study population. BMC Pulm Med. 2009 May 8;9:17. doi: 10.1186/1471-2466-9-17. PMID 19426496
- [Result] Ly NP, Ruiz-Perez B, McLoughlin RM, Visness CM, Wallace PK, Cruikshank WW, Tzianabos AO, O'Connor GT, Gold DR, Gern JE. Characterization of regulatory T cells in urban newborns. Clin Mol Allergy. 2009 Jul 8;7:8. doi: 10.1186/1476-7961-7-8. PMID 19586545
- [Result] Shreffler WG, Visness CM, Burger M, Cruikshank WW, Lederman HM, de la Morena M, Grindle K, Calatroni A, Sampson HA, Gern JE. Standardization and performance evaluation of mononuclear cell cytokine secretion assays in a multicenter study. BMC Immunol. 2006 Dec 12;7:29. doi: 10.1186/1471-2172-7-29. PMID 17156490
- [Result] Gern JE, Calatroni A, Jaffee KF, Lynn H, Dresen A, Cruikshank WW, Lederman HM, Sampson HA, Shreffler W, Bacharier LB, Gergen PJ, Gold DR, Kattan M, O'Connor GT, Sandel MT, Wood RA, Bloomberg GR. Patterns of immune development in urban preschoolers with recurrent wheeze and/or atopy. J Allergy Clin Immunol. 2017 Sep;140(3):836-844.e7. doi: 10.1016/j.jaci.2016.10.052. Epub 2017 Jan 13. PMID 28089873
- [Result] O'Connor GT, Lynch SV, Bloomberg GR, Kattan M, Wood RA, Gergen PJ, Jaffee KF, Calatroni A, Bacharier LB, Beigelman A, Sandel MT, Johnson CC, Faruqi A, Santee C, Fujimura KE, Fadrosh D, Boushey H, Visness CM, Gern JE. Early-life home environment and risk of asthma among inner-city children. J Allergy Clin Immunol. 2018 Apr;141(4):1468-1475. doi: 10.1016/j.jaci.2017.06.040. Epub 2017 Sep 19. PMID 28939248
- [Result] Ramratnam SK, Visness CM, Jaffee KF, Bloomberg GR, Kattan M, Sandel MT, Wood RA, Gern JE, Wright RJ. Relationships among Maternal Stress and Depression, Type 2 Responses, and Recurrent Wheezing at Age 3 Years in Low-Income Urban Families. Am J Respir Crit Care Med. 2017 Mar 1;195(5):674-681. doi: 10.1164/rccm.201602-0272OC. PMID 27654103
- [Result] Kattan M, Bacharier LB, O'Connor GT, Cohen R, Sorkness RL, Morgan W, Gergen PJ, Jaffee KF, Visness CM, Wood RA, Bloomberg GR, Doyle S, Burton R, Gern JE. Spirometry and Impulse Oscillometry in Preschool Children: Acceptability and Relationship to Maternal Smoking in Pregnancy. J Allergy Clin Immunol Pract. 2018 Sep-Oct;6(5):1596-1603.e6. doi: 10.1016/j.jaip.2017.12.028. Epub 2018 Feb 13. PMID 29449165
- [Result] Altman MC, Whalen E, Togias A, O'Connor GT, Bacharier LB, Bloomberg GR, Kattan M, Wood RA, Presnell S, LeBeau P, Jaffee K, Visness CM, Busse WW, Gern JE. Allergen-induced activation of natural killer cells represents an early-life immune response in the development of allergic asthma. J Allergy Clin Immunol. 2018 Dec;142(6):1856-1866. doi: 10.1016/j.jaci.2018.02.019. Epub 2018 Mar 5. PMID 29518416
- [Result] Chandra S, Wingender G, Greenbaum JA, Khurana A, Gholami AM, Ganesan AP, Rosenbach M, Jaffee K, Gern JE, Wood R, O'Connor G, Sandel M, Kattan M, Bacharier L, Togias A, Horner AA, Kronenberg M. Development of Asthma in Inner-City Children: Possible Roles of MAIT Cells and Variation in the Home Environment. J Immunol. 2018 Mar 15;200(6):1995-2003. doi: 10.4049/jimmunol.1701525. Epub 2018 Feb 5. PMID 29431692
- [Result] Bacharier LB, Beigelman A, Calatroni A, Jackson DJ, Gergen PJ, O'Connor GT, Kattan M, Wood RA, Sandel MT, Lynch SV, Fujimura KE, Fadrosh DW, Santee CA, Boushey H, Visness CM, Gern JE; NIAID sponsored Inner-City Asthma Consortium. Longitudinal Phenotypes of Respiratory Health in a High-Risk Urban Birth Cohort. Am J Respir Crit Care Med. 2019 Jan 1;199(1):71-82. doi: 10.1164/rccm.201801-0190OC. PMID 30079758
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT), NIAID — https://www.niaid.nih.gov/about/dait

DOCUMENTS (2):
  • Study Protocol (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT00114881/Prot_000.pdf
  • Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT00114881/ICF_001.pdf